CLINICAL TRIAL: NCT01750814
Title: A Phase III, Randomized, Double-blind, Multi-center Study to Compare the Immunological Efficacy and Safety of GC3102C With GC FLU Inj. Administered Intramuscularly in Healthy Adults
Brief Title: To Evaluate the Effectiveness(Immunogenicity) and Safety of 'GC3102C' Administered Intramuscularly in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GC3102C_P3
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Prophylaxis Against Influenza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GC FLU inj. (Active Comparator): Influneza vaccine, single-dose vial
  Interventions: Biological: GC FLU inj.
- GC3102C (Experimental): Influneza vaccine, multi-dose vial
  Interventions: Biological: GC3102C

INTERVENTIONS:
Biological: GC3102C — a single dose (0.5 mL) intramuscularly on the deltoid muscle
  Arms: GC3102C
Biological: GC FLU inj. — a single dose (0.5 mL) intramuscularly on the deltoid muscle
  Arms: GC FLU inj.

SUMMARY:
The primary objective is to demonstrate the immunological non-inferiority between GC3102C and GC FLU inj. influenza vaccines by assessing geometric mean titers(GMTs) in healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, 18 to <60 years old
* Subjets willing to provide written informed consent and able to comply with the requirements for the study

Exclusion Criteria:

* Subjects with a history of hypersensitivity, especially anaphylactic reactions to egg, egg proteins, chicken or components of vaccine such as gentamicin, gelatin, and arginine
* Subjects with a history of Guillain-Barré syndrome
* Subjects with severe chronic diseases (e.g., cardiovascular diseases without controllable hypertension, hemoglobinopathy, respiratory, metabolic, and renal disorders) who are considered by the investigator to be ineligible for the study
* Subjects previously treated with anti-coagulant therapy or hemophiliac patients who may be at risk of severe hemorrhage after an intramuscular injection
* Subjects who have had an acute febrile (at least 38.0°C) episode at some time during the 72 hours before enrollment
* Subjects who have received a vaccination within 7 days before enrollment or who are scheduled for another vaccination (excluding the study vaccine) during the study
* Immunocompromised subjects with immunodeficiency diseases or those who are receiving immunosuppressive or immunomodulatory therapy, e.g., azathioprine, cyclosporin, interferon, granulocyte-colony stimulating factor, tacrolimus, everolimus, sirolimus
* Subjects who have received high-dose corticosteroids in the 3 months before vaccination or who will be administered a cumulative dose of 700 mg of corticosteroids during the study. Inhaled, intranasal, and local application of corticosteroids is permitted, regardless of dosage, and corticosteroids such as prednisolone at a maximum dose of 15 mg/day are allowed
* Subjects who have been administered immunoglobulins or blood-derived products 3 months before enrollment or who are scheduled for the administration during the study
* Subjects who have received an influenza vaccine within 6 months of enrollment
* A female subject who is pregnant or who is breast-feeding. Subjects of childbearing potential without an appropriate contraceptive measure within 30 days before enrollment and who do not agree to use a clinically acceptable method of birth control during the study (e.g., oral contraceptives, condom, diaphragm or intrauterine device, or vasectomy of male partner)
* Subjects who have participated in any other clinical trials within 30 days of the administration of the study vaccine
* Individuals with other clinically significant medical or psychological condition who are considered by the investigator to be ineligible for the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2013-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
GMT, using the Hemagglutination inhibition(HI) antibody titer | Day 21

SECONDARY OUTCOMES:
Rate of subjects achieving seroconversion | Day 0 , Day 21
Rate of subjects achieving seroprotection | Day 21
Number of Participants Reporting a Solicited Adverse Events After Vaccination | Day 6
Number of Participants Reporting a Unsolicited Adverse Events After Vaccination | Day 21